CLINICAL TRIAL: NCT07097987
Title: Evaluation of the Efficacy of the Composite WM Formula in Promoting GLP-1 Secretion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 25-048-A
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Probiotic; Prebiotic; Glucagon-like peptide-1 (GLP-1); Blood glucose; Insulin
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Arabinose; Erythritol; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control group (Placebo Comparator): Participants in the control group will consume 50 mL water
  Interventions: Other: Control group
- Experimental: WM formula Group (Active Comparator): Participants in the intervention group will consume a single dose of WM formula drink (50 mL) on the study day. The formula includes Bifidobacterium breve (probiotic), ClpB formula (prebiotic), and Rocket Apple extract.
  Interventions: Dietary Supplement: WM formula Group

INTERVENTIONS:
Dietary Supplement: WM formula Group — Participants in the intervention group will consume a single dose of WM formula drink (50 mL) on the study day. The formula includes Bifidobacterium breve (probiotic), ClpB formula (prebiotic), and Rocket Apple extract. The ClpB formula consists of kombucha, soy peptide powder, L-arabinose and erythritol.
  Other Names: Bifidobacterium breve; ClpB formula consists of kombucha, soy peptide powder, L-arabinose and erythritol.; Rocket Apple extract
  Arms: Experimental: WM formula Group
Other: Control group — Participants in the control group will consume 50 mL water
  Arms: No Intervention: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the physiological effects of a WM Formula on glucagon-like peptide-1 (GLP-1) secretion and glycemic regulation in adults with elevated body fat percentage. The WM Formula is a multi-component dietary supplement composed of Bifidobacterium breve (probiotic), ClpB Formula-a prebiotic blend containing probiotic kombucha extract, soy peptide powder, L-arabinose, and erythritol-and rocket apple extract.

Participants enrolled in the study will be required to undergo blood collection, height measurement, body composition analysis, and questionnaire completion. Each testing session will take approximately 5 hours, and participants will need to complete two trial visits in total. There will be a 7-day washout period between the two trial sessions (i.e., after completion of the first trial, the second trial will be scheduled at least 7 days later). On each trial day, blood samples and relevant assessments will be conducted at the following time points: before ingestion of the test product or water, and at 15, 30, 45, 60, 90, 120, and 240 minutes post-ingestion.

DETAILED DESCRIPTION:
This study is a single-center, crossover clinical trial in which each participant serves as their own control. The aim is to evaluate the effects of the WM Formula dietary supplement on promoting endogenous GLP-1 secretion and suppressing appetite in adults with elevated body fat percentage.

Eligible participants will be adults aged 18 years or older, screened based on body fat percentage.

Inclusion criteria:

-Body fat percentage ≥30% for females or ≥25% for males.

Exclusion criteria:

* Prior use of GLP-1 receptor agonists approved in Taiwan (e.g., liraglutide, semaglutide, dulaglutide),
* Use of blood glucose-regulating medications,
* Presence of major organic diseases, Or a history of hypoglycemia.

After enrollment, participants will be required to visit TCI Co., Ltd. for blood collection, height and body composition measurements, and completion of questionnaires. Each study visit will take approximately 5 hours, and participants will undergo two test sessions, separated by a 7-day washout period (i.e., after completing the first test, the second will occur at least 7 days later).

On each test day, blood samples (~14 mL per time point) will be collected via an indwelling venous catheter at the following time points: before ingestion of the test product or water, and at 15, 30, 45, 60, 90, 120, and 240 minutes post-ingestion. The blood samples will be analyzed for GLP-1, DPP-4, complete blood count (CBC), blood glucose, and insulin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older who are willing to sign the informed consent form.
* Body fat percentage: ≥30% for females and ≥25% for males.
* Non-pregnant and non-lactating women who agree to use physical contraceptive methods (e.g., condoms, intrauterine devices) throughout the study period.

Exclusion Criteria:

* Use of GLP-1 receptor agonists approved in Taiwan (e.g., liraglutide, semaglutide, dulaglutide), blood glucose-regulating medications, weight loss-related drugs or functional foods, probiotics, or gastrointestinal health-related supplements or medications within 30 days prior to the start of the study.
* History of chronic gastrointestinal disorders, seizure disorders or epilepsy, hepatic or renal diseases, malignancies, endocrine disorders, psychiatric illnesses, alcohol or drug abuse, or other major organic diseases based on medical history.
* History of gastrointestinal surgery, organ transplantation, or other major surgeries.
* History of hypoglycemia.
* Known lactose intolerance.
* Chronic diarrhea.
* Acute gastroenteritis within 2 weeks prior to study initiation.
* Known allergy to any ingredient in the investigational product.
* Employees or immediate family members of TCI Co., Ltd.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma GLP-1 concentration (pmol/L) | Day 1 and Day 7
  Plasma GLP-1 levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the WM Formula on Days 1 and 7.
Blood glucose concentration (mg/dL) | Day 1 and Day 7
  Blood glucose levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the WM Formula on Days 1 and 7.
Serum insulin concentration (μIU/mL) | Day 1 and Day 7
  Serum insulin levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the WM Formula on Days 1 and 7.
Plasma DPP-4 concentration (ng/mL) | Day 1 and Day 7
  Plasma DPP-4 levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the WM Formula on Days 1 and 7.

CONTACTS AND LOCATIONS:
Locations (1):
- TCI Co., Ltd., Taipei, Taiwan